CLINICAL TRIAL: NCT01559792
Title: Gastric Banding to Bypass - Metabolism Kinetics in Gastric Bypass and Banding
Brief Title: Band to Bypass - Metabolism Kinetics in Gastric Bypass and Banding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Siv Hesse Jacobsen, MD, Hvidovre University Hospital
Other Study IDs: BG092011
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Gastric Bypass; Gastric Banding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators want to study the changes in secretion of gastrointestinal hormones, absorption and metabolism of food and liquids before and after gastric bypass and in patients who are gastric banded but are getting conversion to a gastric bypass. All patients are with normal glucose tolerance. The investigators hypothesis that food uptake/absorption of food is faster after gastric bypass and the secretion of gastrointestinal hormones change.

ELIGIBILITY:
Inclusion Criteria:

* Normal glucose tolerance
* Patients who are undergoing gastric bypass and patients with a gastric band to are converted to gastric bypass

Exclusion Criteria:

* Diabetes,
* Study population must undergo gastric bypass

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all with normal glucose tolerance - patients who are undergoing gastric bypass and patients with a gastric band to are converted to gastric bypass
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Hvidovre
  - Hvidovre hospital, Hvidovre

REFERENCES:
- [Derived] Bojsen-Moller KN, Jacobsen SH, Dirksen C, Jorgensen NB, Reitelseder S, Jensen JE, Kristiansen VB, Holst JJ, van Hall G, Madsbad S. Accelerated protein digestion and amino acid absorption after Roux-en-Y gastric bypass. Am J Clin Nutr. 2015 Sep;102(3):600-7. doi: 10.3945/ajcn.115.109298. Epub 2015 Aug 5. PMID 26245808
- [Derived] Jacobsen SH, Bojsen-Moller KN, Dirksen C, Jorgensen NB, Clausen TR, Wulff BS, Kristiansen VB, Worm D, Hansen DL, Holst JJ, van Hall G, Madsbad S. Effects of gastric bypass surgery on glucose absorption and metabolism during a mixed meal in glucose-tolerant individuals. Diabetologia. 2013 Oct;56(10):2250-4. doi: 10.1007/s00125-013-3003-0. Epub 2013 Jul 27. PMID 23893303